CLINICAL TRIAL: NCT06819826
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of SC0062 Capsule in Patients with IgA Nephropathy and Proteinuria (SUCCESS-1)
Brief Title: A Study of SC0062 Capsule for the Treatment of IgA Nephropathy with Proteinuria
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SC0062-301
Record Dates: First submitted 2025-01-31; First posted 2025-02-11 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: Endothelin Type A Receptor Antagonist
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SC0062 group (Experimental): Subjects will take two capsules daily and the background medication for 108 weeks during the treatment period
  Interventions: Drug: SC0062 strength 10mg
- Placebo group (Placebo Comparator): Subjects will take two capsules daily and the background medication for 108 weeks during the treatment period
  Interventions: Drug: Placebo matched to SC0062

INTERVENTIONS:
Drug: SC0062 strength 10mg — Subjects will take 20 mg once daily for 108 weeks during the treatment period.
  Arms: SC0062 group
Drug: Placebo matched to SC0062 — Subjects will take 20 mg once daily for 108 weeks during the treatment period.
  Arms: Placebo group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase III study to evaluate the efficacy and safety of SC0062 capsule compared to placebo in patients with IgA nephropathy in the presence of proteinuria. The participants must have a high risk of disease progression, despite of stable use of the maximum tolerated labelled or optimized dose of RAASi and/or SGLT2i for at least 12 weeks prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent and fully understand and comply with trial procedures;
* Age ≥18 years old, gender unlimited;
* IgA nephropathy patients with proteinuria must meet all of the following conditions:

  1. According to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI, 2009) creatinine equation, after 12 weeks of the stable use of the background therapy, the mean of two estimated glomerular filtration rates (eGFR) calculated from central laboratory results was ≥ 30 and < 90 mL/min/1.73m2.
  2. Received the maximum labeled or tolerated dose of RAASi (ACEI or ARB) for at least 12 weeks before randomization; If subjects were treated with SGLT2i, MRA, or GLP-1RA prior to randomization, the stable use was also required for at least 12 weeks (maximum tolerated and optimal dose determined by the investigator; Subjects who are intolerant to RAASi may also be enrolled).
  3. The pathological examination confirmed IgA nephropathy. Two 24-hour urine samples were collected during the screening period, after 12 weeks of the stable use of the background treatment. Both of the results conducted by the central laboratory were met: 24-hour urine protein to creatinine ratio (UPCR) ≥ 0.75 g/g or 24-hour urinary protein excretion rate (UPER) ≥ 1.0 g.
* Laboratory tests shall meet the following criteria:

  1. Serum albumin ≥ 30 g/L;
  2. Hemoglobin ≥ 90 g/L ; Platelet count ≥80×109/L;
  3. Brain natriuretic peptide (BNP) ≤ 200 pg/mL or N-terminal pro B-type natriuretic peptide (NT-proBNP) ≤ 600 pg/mL;
  4. Blood potassium ≤ 5.5 mmol/L;
  5. Systolic blood pressure (SBP) ≤ 160 mmHg;
  6. Hemoglobin A1c ≤ 8%;
  7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2×ULN; Total bilirubin ≤ 1.5×ULN;
* During the entire study period from the signing of the informed consent to 3 months after the final administration, fertile females and males who have not received vasectomy should take effective contraceptive measures [Effective contraceptive measures include: Vasectomy, intrauterine device (IUD), hormones (oral, patch, ring, injection, implant) and barrier methods (diaphragm, cervical cap, sponge, condom).

Exclusion Criteria:

* Pregnant or lactating females; Women of childbearing potential (WOCBP) who have a positive blood pregnancy test before randomization;
* A history of hypersensitivity or allergic to any component of the study drug (SC0062 capsule);
* Systemic use of corticosteroids or immunosuppressants for more than 2 weeks within 3 months prior to randomization; The following are excluded: local topical or intraarticular, intranasal and inhaled glucocorticoids; Use of biological agents (such as rituximab, Telitacicept, etc.), Iptacopan capsules, budesonide enteric-coated capsules within 6 months prior to randomization;
* Concurrent diagnosis of chronic kidney disease caused by other etiologies (including polycystic kidney disease, diabetic kidney disease, or other primary glomerular disease) as determined by the investigator;
* Secondary IgA nephropathy, including but not limited to: Henoch-Schönlein purpura, ankylosing spondylitis, systemic lupus erythematosus, amyloidosis, etc.
* Renal biopsy results showed that > 25% of glomeruli with crescents, or interstitial fibrosis/tubular atrophy > 50%;
* Based on KDIGO guidelines, rapidly progressive glomerulonephritis was clinically suspected (judged by the investigator);
* Nephrotic syndrome (UPER > 3.5g/d and serum albumin < 30g/L, with or without edema and hyperlipidemia) at screening;
* A history of any lung disease requiring oxygen therapy (e.g., chronic obstructive pulmonary disease, emphysema, pulmonary edema, etc.);
* Use of the same class drug (endothelin receptor antagonist, ERA) before randomization;
* A history of moderate or severe edema, non-traumatic facial edema, or myxedema within the 6 months prior to randomization;
* A history of orthostatic hypotension within 6 months before randomization;
* A history of clinically significant cirrhosis assessed by the investigator;
* A history of worsening heart failure, acute coronary syndrome, transient ischemic attack, stroke and other serious cardiovascular and cerebrovascular diseases within 6 months prior to randomization, or NYHA Grade III to IV at screening;
* A history of kidney or other organ transplantation (except corneal transplantation);
* A condition which had the potential to interfere with oral drug absorption, such as subtotal gastrectomy, clinically severe gastrointestinal disorders, or certain types of bariatric surgery;
* Use of potent CYP3A4 inducers and potent CYP3A4 inhibitors within 2 weeks (14 days) before randomization;
* Received other treatment for IgA nephropathy within 28 days prior to randomization except as permitted by the protocol;
* Active Hepatitis B, active Hepatitis C, active syphilis and Hiv-positive ;
* A history of malignant tumors within 5 years, except for skin squamous cell carcinoma, colon polyp or in situ cervical cancer, thyroid papillary carcinoma;
* A history of alcohol or drug abuse or dependence, or a history of mental illness;
* Participated in clinical trials of other investigational drugs or medical devices within 3 months prior to randomization;
* Any other clinically significant disease, condition, or medical history that may interfere with subjects' safety, study evaluation, and/or study procedures at the discretion of the investigator;
* Any other reasons for not being suitable for participating in this clinical study at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-02-14 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour urine protein-to-creatinine ratio (24h-UPCR) at 36 weeks | Baseline, 36 weeks
  UPCR is measured from the 24-hour urine collection samples.

SECONDARY OUTCOMES:
Change from baseline in estimated glomerular filtration rate (eGFR) at 108 weeks | Baseline, 108 weeks
  Estimated glomerular filtration rate (eGFR) will be calculated based on the 2009 CKD-EPI equation.
The total slope of estimated glomerular filtration rate (eGFR) from baseline to 108 weeks | Each visit from baseline to 108 weeks
  the total eGFR slope is defined as the mean rate of change in eGFR from baseline to 108 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Yuexiu District, China